CLINICAL TRIAL: NCT05641857
Title: Lumbar Spine on MRI and Low Back Pain in Elite Cross-country Skiers
Status: Completed | Type: Observational
Sponsor: Orton Orthopaedic Hospital (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other); Päijät Häme Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 465
Record Dates: First submitted 2022-11-29; First posted 2022-12-08 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Disc Degeneration
Keywords: low back pain; disc degeneration; athlete; matched case control
MeSH Terms: conditions — Intervertebral Disc Degeneration; Low Back Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low back pain and disc degeneration among elite cross-country skiers: No intervention Interview, clinical examination and MRI
- Low back pain and disc degeneration among healthy volunteers: No intervention Interview, clinical examination and MRI

SUMMARY:
The investigators will examine the prevalence of low-back pain and disc degeneration among Finnish elite skiers between 16 and 35 years of age and compare these findings with the data collected among healthy volunteers studied between 1994-2021.

DETAILED DESCRIPTION:
The study population will consist of Finnish elite cross-country skiers between 18 and 35 years of age. Invitation letters will be sent to all skiers who are selected to national teams at season 2022-2023. The study population for the current study will be approximately 100 individuals. Study protocol for the current study will consist of a semi-structured interview, clinical examination, lumbar spine MRI and patient reported outcome measures. All participants will sign an informed consent before commencement of the study. If a participant is younger than 18 years, also his/her caregiver will be asked for a signed consent.

The interview comprised of questions about the athletes training volume and possible LBP without associated trauma. (suspension from training or competition due to LBP, possible contacts to health-care providers).

Body height and weight were self-reported. Leg length inequality was assessed comparing the height of the left and right iliac crests in standing position with straight knees. Wooden blocks of different thickness (with 0.5 cm increment) were used for correction of possible leg length inequality. Symmetry of the back was measured in forward bending using a scoliometer.

From MRI (high field 1.5 T) the signal intensity of the nucleus pulposus will be assessed both qualitatively and quantitatively. The midline T2-weighted images will be independently evaluated visually by three evaluators using a Pfirrmann classification. The quantitative nucleus signal intensities will be assessed by two evaluators using a relative measure comparing the signal intensity of the nucleus pulposus to that of the adjacent cerebrospinal fluid on T2-weighted images.

ELIGIBILITY:
Inclusion Criteria:

* Finnish elite cross-country skiers (national teams from the age of 16)

Exclusion Criteria:

* none

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All skiers who are selected to the national teams at season 2022-2023.
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Pfirrmann summary score | Baseline
  Summary score of individual Pfirrmann grades of lumbar discs (L1-L5). Grade is 5 to 25, where 5 is the best value and 25 the worst value.
Low back pain (LBP) | Baseline
  Low back pain NRS (numeric rating scale) 0 to 10, where 0 is the best value and 100 is the worst value.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) | Baseline
  Oswestry Disability Index, 0 to 100, where 0 is the best value and 100 the worst value.
EQ-5D-5L | Baseline
  The health-related quality of life, 0 to 100, where 0 is the worst value and 100 the best value.

CONTACTS AND LOCATIONS:
Overall Officials: Teija Lund, Study Director — Helsinki University Hospital and Helsinki University; Anni Aavikko, Principal Investigator — PHHYKY
Locations (1):
- Research Institute Orton, Helsinki, In the USA Or Canada, Please Select..., Finland

REFERENCES:
- [Derived] Aavikko A, Pesonen J, Ristolainen L, Murto N, Kautiainen H, Lund T. Prevalence of Low Back Pain and Disc Degeneration in Elite Cross-Country Skiers: A Comparative Study With Non-Athlete Controls. Scand J Med Sci Sports. 2025 Dec;35(12):e70187. doi: 10.1111/sms.70187. PMID 41416933